CLINICAL TRIAL: NCT04095000
Title: Health Equity: Advance Care Planning for Spanish Speaking Teens With Cancer-1st Resubmission
Acronym: FACE-TC-Sp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maureen Lyon (Other)
Responsible Party: Sponsor-Investigator, Maureen Lyon, Professor of Pediatrics, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB 11473
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This pilot will use a randomized control trial (RCT) design with the intent to treat. Randomization will be generated by computer to ensure the same numbers will be recruited to the FACE-TC Sp intervention and Treatment As Usual comparison group without bias, using a 1:1 ratio. We estimate that 32 adolescents ever diagnosed with cancer, aged 14 to 21, and 32 guardians/surrogates (N=64) will be enrolled and receive secondary screening. They will complete a Demographic Data Sheet. The assent/consent process focuses on readiness to participate, potential barriers to participation, as well as enhancing motivation. Adolescents and families will then be screened for eligibility. Eligible dyads, estimated to be 30 dyads, will complete baseline data. Then, the adolescent/family dyad will be randomly assigned to one of two conditions: 15 dyads will be assigned to FACE-TC SP and 15 dyads to Treatment As Usual.
Who Masked: Outcomes Assessor
Masking Description: RA-Assessor will be blinded to randomization to reduce bias in collecting questionnaire data and data abstraction from electronic health record.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FACE-TC SP (Experimental): The current FACE-TC protocol consists of three weekly 60 to 90-minute sessions in a dyadic format facilitated by a trained/certified interviewer. If our community partners recommend otherwise, this structure could change. Each session is followed by a 10-minute assessment, using process measures to assess participants' ratings of the quality of communication and satisfaction.
  Interventions: Behavioral: FACE-TC SP
- Treatment As Usual (Active Comparator): Treatment as Usual comparison condition will also be assessed and measures administered at the same time intervals.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: FACE-TC SP — The current FACE-TC protocol consists of three weekly 60 to 90-minute sessions in a dyadic format facilitated by a trained/certified interviewer. If our community partners recommend otherwise, this structure could change. Each session is followed by a 10-minute assessment, using process measures to assess participants' ratings of the quality of communication and satisfaction.
  Arms: FACE-TC SP
Behavioral: Treatment as Usual — Treatment as Usual comparison condition will also be assessed and measures administered at the same time intervals.
  Arms: Treatment As Usual

SUMMARY:
Pediatric ACP (Advance Care Planning) (pACP) (1) Supports communication with children/adolescents at any stage of a serious illness in understanding their illness, complications, fears, and hopes, as well as treatment preferences regarding future medical care with their family; (2) Communicates these goals of care and treatment preferences with their physician; and (3) Documents these goals of care and end-of-life treatment preferences. Among adolescents, cancer is the leading cause of disease-related deaths. Survival has improved far less for 15 to 24 year-olds than it has for older patients. About one-fourth will die prematurely. No pediatric Advance Care Planning (pACP) model exists to serve Spanish speaking adolescents with cancer.

Objective: To take first steps to implement pACP as a routine, structured intervention in pediatric hospitals with underserved Spanish speaking adolescents living with cancer through timely conversations with their families to relieve suffering (physical, psychological, spiritual) and maximize the quality of life

DETAILED DESCRIPTION:
Non-English-speaking patients are far less likely to have advance care planning documents than English speakers. Some ethnicities in an adult study had no patients with an advance care planning document. Since completing advance care planning may increase early palliative care enrollment, as it did in the FACE-TC study, strategies to promote pACP are urgently needed, particularly with non-English speaking patients.

Transactional stress and coping theory is the basis for the FACE intervention, because interventions can change the appraisal of an illness from that of a death threat to a challenge with potential for personal growth and mastery.

Many adolescents want to talk about their goals and values regarding their own end-of-life care. These important discussions are often regarded as needed, but not initiated before a medical crisis, due to perceived (and unwarranted) fears they will cause anxiety, take away hope or cause physician or family discomfort. Parents who discussed death with their children who were dying of cancer reported no regrets. Pediatric ACP for adolescent cancer patients is a public health issue, because of its high burden and potential for the prevention of suffering, as most teen and young adult cancer patients at end of life get aggressive care. The proposed study will explore prospectively whether Hispanic/Latino teens can be safely supported to help them make informed choices with their families, advancing clinical practice. Heretofore, family refers to the legal guardian(s) or surrogate decision maker(s) of the adolescent patient with cancer.

Age appropriate communication that includes the adolescent and family can facilitate decisions about medical treatments that precede death. Competency to participate in decision-making has been challenged by research on adolescent brain development, which demonstrates the structure of the adolescent brain is not fully formed.

However, what these findings mean in terms of the actual functioning or behavior of an individual adolescent is unclear, stirring up legal and public policy debates. The implications for pACP are unclear. Empirical evidence and the ethical principles of justice and autonomy support the practice of including adolescents in decision-making about their future medical care, if they could not speak for themselves. Cognitive capacities required for "informed consent" for medical treatment exist in early adolescence. Nor is there reason to suspect that young adolescents have a less mature understanding of death: irreversibility; finality or non-functionality; universality or inevitability; and causality. Hinds and colleagues found that children with cancer realized they were involved in an end-of-life decision, understood the consequences of their decision (that death is the outcome no matter what), and could share the reasons for their preferences. The decision factors most frequently reported by pediatric patients were relationship based, while parents identified good communication. Parents also thought that communicating with the child about end-of-life preferences was appropriate when approached with sensitivity and care. The issues facing adolescents with a life-threatening illness are different from those facing adults, because minors' preferences are not legally binding.

Culture and ethnicity are important in pACP. Cultural values differ with respect to patient autonomy. For those adolescents who do not want to defer these decisions to their family or physician, culturally sensitive pACP conversations may ensure patients and families feel cared for and supported, when there is full participation by the family and clear communication to the physician. Hospice surveys show one-third of Latinos opposed life support that prolonged suffering, leading the National Hospice and Palliative Care Organization to actively reach out to Latino communities. Immigrant status influences decisions about aggressive treatments, suggesting there may not be disparities in EOL care, but rather differences in preferences. Investigators will explore whether the number of years residing in the U.S. influences treatment choices among study participants.

The FACE intervention is informed by the American Academy of Pediatrics, the Institute of Medicine (IOM), institutional guidelines, and evolving practice and theory recommending: (1) that decisions about end-of-life (EOL) care be shared among the adolescent patient, family, and physician; (2) that these discussions take place when the patient is stable; (3) and that decisions be individualized. In the SUPPORT study physicians misunderstood the patient's preferences about CPR in 80% of the cases. Clinical reports suggest that parents and physicians sometimes disregard adolescents' previously expressed wishes, particularly with regard to forgoing life-sustaining treatment. One of the goals of this intervention is to increase the congruence in treatment preferences between Spanish speaking adolescents with cancer and their families. Investigators also hope to resolve potential conflict about these decisions within the structure of the intervention through referrals to the ethics committee and chaplaincy program. One way the proposed FACE-TC Sp intervention differs from the SUPPORT study is that investigators include both the patient and surrogate in the decision-making process by actively engaging interested adolescents and families in facilitated conversations by a highly trained/certified interviewer about the end-of-life preferences that adolescents have.

Only three pediatric ACP (pACP) programs are reported in the peer reviewed literature.1 A qualitative study, FOOTPRINTS™, focused on patients aged 8-20 years with Duchennes' Muscular Dystrophy. The second involved conversations between an ethicist and parents of children who were dying about the parent's goals for their child's care. Voicing My CHOICES™ is a model currently being tested with young adults by Wiener and colleagues. Investigators are exploring whether completion of an ACP document, by seriously ill young adults will foster future discussions with family and the physician regarding the young adult's personal goals, values or beliefs. Only Lyon's (PI) pilot study of FAmily CEntered ACP for Teens with Cancer (FACE-TC) employed a randomized controlled trial (RCT) to evaluate a structured pACP intervention. Adolescents/family dyads were randomized to FACE-TC Sp or a Treatment as Usual condition. See Preliminary Studies. In a systematic review of children's engagement in health related decisions, only the FACE pilot focused on children's participation in decisions about their medical care with their family. The FACE pACP approach offers the following advantages over other previous approaches. It is family-centered and disease-specific. It integrates the Representational Approach to Patient Education, which focuses first on assisting individuals to understand their medical condition, to explore values and goals, and to begin weighing the benefits and burdens of any life-sustaining treatment compared to personal/family values and goals. It is delivered by trained/certified facilitators. It focuses on promoting psychological well-being in the face of serious illness, consistent with the recommendations of Folkman. This inclusion of families is a core value of Spanish speaking families, as is religion. A majority of Hispanic adults (55%) say they are Catholic, while 16% are evangelical Protestants and 5% are mainline Protestants.

The adaptation and pilot test of FACE-TC Sp will advance scientific knowledge by contributing to understanding what Hispanic/Latino adolescents living with cancer want with respect to goals of care and treatment preferences in the context of family support and enable us to put into practice recommended policies and understand how culture and spiritual experiences influence pACP outcomes.

ELIGIBILITY:
Adolescent Inclusion Criteria:

* ≥14.0 years and <21.0 years at the time of enrollment
* primary language is Spanish

Surrogate Inclusion Criteria:

* >17 years

Exclusion Criteria for adolescents and surrogate decision makers/legal guardians:

* currently experiencing symptoms of depression in the severe range, homicidality, suicidality or psychosis at secondary screening
* known to be developmentally delayed

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-08-05 (Actual); Study Completion 2021-08-05 (Actual)

PRIMARY OUTCOMES:
Development/Adaptation FACE TC for Spanish Speaking Teens | 6 months
  Adapting and tailoring this evidence-based intervention will be accomplished through well-established techniques. The community partner interviews will be achieved through our youth with cancer, families affected by cancer and community stakeholders. Logic modeling based on our previous research and a literature review is completed.
  Study 1: Adolescent Focus Group: Do Hispanic/Latino Adolescents and Families Want to Be Involved in pediatric Advance Care Planning? We will conduct a 60 minute audio-taped focus group with five teens with cancer, ages 14-17, regarding what they would want and need when it comes to EOL care, as we have with our previous adaptations/development.11,59 We will review the English speaking version of the FACE protocol for changes (e.g. number of sessions, Five Wishes vs. Voicing My Choices).
Lyon Advance Care Planning Survey-Adolescent & Family Versions | 6 months
  With the assistance of Children's National's Language Services (See Letter of Support) and our Hispanic chaplain and research staff we will translate and back translate the Lyon Advance Care Planning Survey-Adolescent and Surrogate version. We will then meet with adolescents with cancer and families to adapt/revise the survey (e.g. number of questions, best way to ask question, reading level).
Family Focus Group with Hispanic/Latino Families about Program Development | 6 months
  Hispanic/Latino family members will be drawn from the Children's National Patient and Family Advisory Council (PFAC). We will conduct a 60 minute audio-taped focus group with Spanish speaking members. How should FACE-TC be adapted so as to be respectful of linguistic and cultural differences?
Critical Review of Revised Protocol | 6 months
  Our community partners will meet in a Science Café to review the revised/adapted FACE-TC SP protocol. Rev. Roque will introduce the issues and the adapted study. We will explore thoughts, feelings and reactions until no new themes emerge and consensus is achieved.

SECONDARY OUTCOMES:
Pilot Test FACE-TC Spanish (FACE-TC Sp) | 24 months
  We are proposing to 1) study the feasibility, acceptability and safety of FACE-TC Sp; and 2) assess the effect of FACE-TC Sp on the primary (congruence in treatment preferences & quality of communication) and secondary outcomes (quality of life & plans and actions). We expect the FACE-TC Sp protocol will offer advantages over the existing standards, where adolescents 18 years of age or over are handed an advance directive form in the emergency department by a clerk or nurse, or otherwise mailed a form on their 18th birthday.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Lyon, PhD, Principal Investigator — Center for Translational Research/Children's Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared. Deidentified data will be shared by contacting the PI upon completion of the study for appropriate research services.

REFERENCES:
- [Result] Lyon ME, Arem H, Jacobs S. Health disparities: Barriers to building effective palliative end-of-life care for Spanish speaking teens with cancer. Clinical Practice in Pediatric Psychology. CPP-2020-0439R1. In press.